CLINICAL TRIAL: NCT03019848
Title: Effect of Oral Supplementation With Curcumin in Patients With Proteinuric Diabetic Kidney Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Magdalena Madero, MD, Chief of the Nephrology Department, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INC.12-793
Record Dates: First submitted 2016-09-12; First posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2016-09

CONDITIONS: Proteinuria
Keywords: Redox and pro-inflammatory status
MeSH Terms: conditions — Proteinuria | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Curcumin (Experimental): Each patient of this group will receive 1.67 grams of curcumin ( 7 capsules of 231 mg) divided in 3 doses daily for 6 months.
  Interventions: Dietary Supplement: Curcumin
- Placebo (Placebo Comparator): The control group will receive 7-capsules/ day identical in color and size, containing placebo for 6 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Curcumin
  Other Names: Tumeric
  Arms: Curcumin
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if the oral supplementation with curcumin reduces proteinuria, improves the redox and pro-inflammatory state in patients with chronic kidney disease associated to Diabetes mellitus.

DETAILED DESCRIPTION:
Diabetic Kidney Disease (DKD) represents the fist cause of end-stage kidney disease in Mexico and the world, and it is characterized by the presence of hyperfiltration, glomerular hypertrophy, tubular albuminuria and mesangial matrix expansion, mainly by the oxidative stress and the pro-inflammatory state.

Current treatments are limited on controlling proteinuria and delay progression of the disease, but even with an optimal management, a significant number of patient progress to end-stage renal disease.

Curcumin, found in the extracts of the rhizome of the plant Curcuma longa L., has a wide spectrum of biological and pharmacological activities, such as anti-oxidant, anti-inflammatory, anti-carcinogenic and anti-diabetic effects. It has the capacity to act directly with highly reactive oxygen species, induce the expression of various cytoprotective proteins through Keap1/Nrf2/ARE pathway and reducing inflammatory transcription factors such as NF-κB and TNF-α.

Curcumin could be an adjuvant treatment in the management of DKC due to his pleiotropic nature, low cost and few side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Diabetes Mellitus type 2 and proteinuric kidney disease with 1000 mg of more proteins in daily recollection
* Glomerular filtration rate between 15-60 mL/min/ 1.73 m2 calculated by CKD-EPI
* Patients taking Angiotensin II Receptor Blocker or ACE inhibitors

Exclusion Criteria:

* Renal replacement therapy
* Autoimmune disease or malignancy
* Pregnancy
* Hepatic damage
* Congestive heart failure classification III or IV (NYHA)
* History of organ transplantation
* History of chemotherapy or immunosuppression within 2 years prior to screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Urine protein excretion | 24 weeks
  Quantify proteinuria and adjust based in creatinuria, before and after the treatment. ( Units: g/g).

SECONDARY OUTCOMES:
Free radical scavenging activity | 6 months
  Free radical scavenging activity in plasma using DPPH, a purple-colored stable free radical is reduced to the yellow-colored diphenyl picryl-hydrazine, and the absorbance will be measure at 518 nm.
  The results were expressed as percentage of DPPH inhibition.
Malondialdehyde (MDA) | 6 months
  Malondialdehyde (MDA) in plasma. We will measure the reaction with 1-methyl-2- phenylindole at 586 nm, using a standard curve of tetrame- thoxypropane.
Proinflammatory status | 6 months
  Enzyme-linked immunoassay (ELISA) will be use to the measurement of serum TGF-b, IL-10, IL-6 and TNF-a.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Cardiologia Ignacio Chávez, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Background] de Zeeuw D, Remuzzi G, Parving HH, Keane WF, Zhang Z, Shahinfar S, Snapinn S, Cooper ME, Mitch WE, Brenner BM. Proteinuria, a target for renoprotection in patients with type 2 diabetic nephropathy: lessons from RENAAL. Kidney Int. 2004 Jun;65(6):2309-20. doi: 10.1111/j.1523-1755.2004.00653.x. PMID 15149345
- [Background] Trujillo J, Chirino YI, Molina-Jijon E, Anderica-Romero AC, Tapia E, Pedraza-Chaverri J. Renoprotective effect of the antioxidant curcumin: Recent findings. Redox Biol. 2013 Sep 17;1(1):448-56. doi: 10.1016/j.redox.2013.09.003. PMID 24191240
- [Background] Khajehdehi P, Pakfetrat M, Javidnia K, Azad F, Malekmakan L, Nasab MH, Dehghanzadeh G. Oral supplementation of turmeric attenuates proteinuria, transforming growth factor-beta and interleukin-8 levels in patients with overt type 2 diabetic nephropathy: a randomized, double-blind and placebo-controlled study. Scand J Urol Nephrol. 2011 Nov;45(5):365-70. doi: 10.3109/00365599.2011.585622. Epub 2011 May 31. PMID 21627399
- [Background] Jimenez-Osorio AS, Garcia-Nino WR, Gonzalez-Reyes S, Alvarez-Mejia AE, Guerra-Leon S, Salazar-Segovia J, Falcon I, Montes de Oca-Solano H, Madero M, Pedraza-Chaverri J. The Effect of Dietary Supplementation With Curcumin on Redox Status and Nrf2 Activation in Patients With Nondiabetic or Diabetic Proteinuric Chronic Kidney Disease: A Pilot Study. J Ren Nutr. 2016 Jul;26(4):237-44. doi: 10.1053/j.jrn.2016.01.013. Epub 2016 Feb 22. PMID 26915483